CLINICAL TRIAL: NCT05075369
Title: Correlation Between Water Drinking Test Study and Disc Hemorrhages in Normal Tension Glaucoma
Brief Title: Water Drinking Test Study and Disc Hemorrhages in Normal Tension Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Lisa Gould, Lisa Gould Associate Professor, University of Manitoba
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: B2021 060; Karla Zuniga (Other: UManitoba)
Record Dates: First submitted 2021-09-19; First posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Normal Tension Glaucoma
Keywords: normal tension glaucoma; disc hemorrhages; water drinking test
MeSH Terms: conditions — Low Tension Glaucoma

STUDY DESIGN:
Intervention Model Description: patients with a diagnosis of normal tension glaucoma and noted to have a disc hemorrhage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- baseline Intraocular pressure (No Intervention): The participants will have their intraocular pressure measured with Goldmann Application Tonometry immediately prior to beginning the water drinking test.
- Change in Intraocular pressure with Water drinking test (Active Comparator): The participants will undergo the water drinking test as previously described, i.e. after drinking 800 mls of water over a 5 minute period, the intraocular pressure will be measured immediately after completion of ingestion, followed by intraocular pressure measurements every 15 minutes for 60 minutes, using etc Goldmann apllantion tonometer.
  Interventions: Diagnostic Test: water drinking test

INTERVENTIONS:
Diagnostic Test: water drinking test — Water drinking test-glaucoma diagnostic test - marker for outflow facility reserve to detect IOP instability when the body ingests 800 ml of water within a 5 minute period of time
  Arms: Change in Intraocular pressure with Water drinking test

SUMMARY:
Disc hemorrhages are a known risk factor for progression of glaucoma. A positive water drinking test is also associated with progression of primary open glaucoma. The purpose of this study is to determine if patients with normal tension glaucoma and disc hemorrhages have a positive water drinking test.

Patients with normal tension glaucoma and a disc hemorrhage will be recruited to undergo a water drinking test prior to any change in their treatment.

DETAILED DESCRIPTION:
Patient with normal tension glaucoma under the care of a fellowship trained glaucoma specialist and noted to have a disc hemorrhage in one or both eyes when examined in the office will be recruited to undergo a water drinking test (WDT). After an informed consent is obtained, arrangements will be made to undergo the WDT either at the ophthalmologist's office or the local hospital clinic(Misericordia). The test will be administered in the following way:

Upon arrival the patients baseline intraocular pressure (IOP) will be measured, then shortly afterwards the patient will drink 800 ml of water in a period of 5 minutes. Immediately after the water ingestion has finished a second IOP will be measured, followed by IOP measurements every 15 minutes for 60 minutes with a Goldman applanation tonometer by the same examiner. All of these measurements will be collected in a data sheet for the WTD. A total of 60 minutes would be the duration of the activity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of normal tension glaucoma by a fellowship trained glaucoma specialist,
* Clinical diagnosis of a disc hemorrhage diagnosed by a fellowship trained glaucoma specialist,
* Must be able to swallow water
* Must be able to be positioned to allow accurate measurement of the Intraocular pressure with a slit lamp mounted Goldmann applanation tonometer
* Must have a smooth corneal surface to allow for accurate Goldmann application tonometry measurement
* Outpatient
* A sufficient level of education to understand study procedures and be able to communicate with site personnel

Exclusion Criteria:

* History of refractive surgery,
* Active ocular infection,
* Pregnancy,
* Cardiac or renal diseases, history of urinary retention,
* Corneal abnormalities preventing reliable IOP measurements,
* Previous trabeculectomy or glaucoma shunt surgery,
* Previous laser iridotomy,
* Cognitive impairment or language barrier preventing ability to provide an informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Change in baseline intraocular pressure(IOP) with water drinking test | The water drinking test takes 60 minutes, and the participant is then finished and can leave.
  The change in intraocular pressure in patients with normal tension glaucoma and a disc hemorrhage after undergoing the water drinking test will be measured with Goldmann applanation tonometry. A change from baseline IOP of 5 mm Hg is considered abnormal .

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Gould, MD FRCS, Principal Investigator — University of Manitoba

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the paper or poster , after deidentification (text, tables, figures, and appendices) will be available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately upon publication and for 36 months afterwards
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Background] Susanna R Jr, Vessani RM, Sakata L, Zacarias LC, Hatanaka M. The relation between intraocular pressure peak in the water drinking test and visual field progression in glaucoma. Br J Ophthalmol. 2005 Oct;89(10):1298-301. doi: 10.1136/bjo.2005.070649. PMID 16170120
- [Background] Susanna R Jr, Clement C, Goldberg I, Hatanaka M. Applications of the water drinking test in glaucoma management. Clin Exp Ophthalmol. 2017 Aug;45(6):625-631. doi: 10.1111/ceo.12925. Epub 2017 Mar 9. PMID 28164419
- [Background] Ishida K, Yamamoto T, Sugiyama K, Kitazawa Y. Disk hemorrhage is a significantly negative prognostic factor in normal-tension glaucoma. Am J Ophthalmol. 2000 Jun;129(6):707-14. doi: 10.1016/s0002-9394(00)00441-4. PMID 10926977